CLINICAL TRIAL: NCT03209843
Title: Post-stenting Assessment of Reendothelialization With OFDI After CTO Procedure
Brief Title: Post-stenting Assessment of Reendothelialization With OFDI After CTO Procedure (PERFECTO)
Acronym: PERFECTO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PERFECTO
Record Dates: First submitted 2017-06-20; First posted 2017-07-06 (Actual); Last update posted 2021-04-14 (Actual); Status verified 2021-04

CONDITIONS: Chronic Total Occlusion of Coronary Artery; Optical Coherence Tomography; Ischemic Cardiomyopathy; Neointimal Hyperplasia; Stent Thrombosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Successfully CTO recanalization (Other)
  Interventions: Procedure: Percutaneous recanalization of chronic total occlusion

INTERVENTIONS:
Procedure: Percutaneous recanalization of chronic total occlusion — Percutaneous recanalization of chronic total occlusion followed by immediate systematic coronary optical frequency domain imaging (OFDI) at inclusion. Intra-individual post stenting assessment of reendothelialization with a second coronary angiography with OFDI analysis at 3 months.

SUMMARY:
The objective of PERFECTO is to assess the reendothelialization at 3 months after successfully CTO percutaneous intervention (PCI) with new generation drug eluting stent (DES) by OFDI analysis. Designed as a multicentric, observational and prospective study which will be conducted at University Hospital of Poitiers (France), a systematic OFDI analysis will be realized immediately after CTO-PCI and at 3 months. Known as major predictive factors of stent thrombosis, percentages of malapposition, uncovered struts and neointimal hyperplasia proliferation will be measured over the entire length of each stent implanted combining in a composite primary endpoint.

ELIGIBILITY:
Inclusion Criteria:

* Successfully CTO revascularization by PCI with immediate post-PCI OFDI analysis
* 3 months follow-up with OFDI analysis of the recanalized coronary artery
* Aged 18 or over
* Written informed consent

Exclusion Criteria:

* Contraindication or impossibility to realize a safety coronary OFDI (severe tortuosities)
* Severe renal insufficiency (creatinine clearance < 30 ml/min)
* Pregnancy or women with child-bearing potential
* Bacteriemia or septicemia
* Severe hemodynamic instability
* Severe coagulation disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2018-03-07 (Actual); Primary Completion 2021-02-12 (Actual); Study Completion 2021-02-12 (Actual)

PRIMARY OUTCOMES:
Percentage of uncovered stent struts | 3 months
  Measured by OFDI 3 months after CTO recanalization every millimeter over entire length of each stent implanted. (Number uncovered struts x 100)/total number of struts.
Percentage of malapposed stent struts | 3 months
  Measured by OFDI 3 months after CTO recanalization every millimeter over entire length of each stent implanted. (Number of malapposed struts x 100)/total number of struts.
Percentage of neointimal hyperplasia proliferation | 3 months
  Measured by OFDI 3 months after CTO recanalization every millimeter over entire length of each stent implanted. [(minimal stent area - minimal lumen area)/minimal stent area]x100.
Minimal lumen area | 3 months
  Measured by OFDI 3 months after CTO recanalization every millimeter over entire length of each stent implanted.
Minimal lumen diameter | 3 months
  Measured by OFDI 3 months after CTO recanalization every millimeter over entire length of each stent implanted
Thrombus | 3 months
  Measured by OFDI 3 months after CTO recanalization every millimeter over entire length of each stent implanted.
Edge dissection | 3 months
  Measured by OFDI 3 months after CTO recanalization every millimeter over entire length of each stent implanted.

SECONDARY OUTCOMES:
Relevancy of immediate post-PCI OFDI analysis | Day one
  To estimate the percentage of patients in whom the post-stenting OFDI analysis will reveal a suboptimal result of angioplasty whereas final angiography was considered optimal, as assessed by the presence of one or more of the following criteria:
  1. Dissection or thrombus.
  2. Residual stenosis.
  3. Stent malapposition defined by at least one malapposed strut.
  4. Residual stenosis.
Impact of the technique employed for CTO revascularization on the reendothelialization | 3 months
  Comparison of primary composite endpoint between different way of recanalization:
  1. Anterograde.
  2. Retrograde.
  3. Dissection/re-entry.
One year clinical follow-up | One year
  Each participating center will perform one year after CTO PCI a clinical evaluation of all patients included. This could be established directly with the subject during medical follow-up or indirectly via family doctor. Standardized questionnaire will be provided at the end of the e-case report form (CRF). Occurrence of major adverse cardiac events (myocardial infarction, death, stroke), sudden death, hospitalization for cardiac disease and severe hemorrhage will be recorded. Any new coronary arteriography will be noticed, as well as any PCI or coronary artery bypass graft (CABG) during this one-year follow-up.
  1. Death all-cause
  2. Myocardial infarction
  3. Stroke
  4. Sudden death
  5. Hospitalization for cardiac cause
  6. Severe hemorrhage
Angina | One year
  About symptoms, the Canadian Cardiovascular Society (CCS) grading system and New York Heart Association functional classification will be used to assess respectively exertion-induced angina and dyspnea, and compared to symptoms recorded before CTO revascularization.
Dyspnea | One year
  About symptoms, the Canadian Cardiovascular Society (CCS) grading system and New York Heart Association functional classification will be used to assess respectively exertion-induced angina and dyspnea, and compared to symptoms recorded before CTO revascularization.

CONTACTS AND LOCATIONS:
Overall Officials: Sebastien Levesque, MD, Principal Investigator — University Hospital of Poitiers, Department of Cardiology
Locations (7):
- France (7):
  - CHU de Clermont-Ferrand, Clermont-Ferrand
  - GHM de Grenoble, Grenoble
  - Bressollette, Nantes
  - CHU de Nimes, Nîmes
  - CHU Poitiers, Poitiers
  - Institut A.Tzanck, Saint-Laurent-du-Var
  - CHU de Toulouse, Toulouse

REFERENCES:
- [Derived] Levesque S, Faurie B, Lattuca B, Lemoine J, Pitchecanin G, Motreff P, Bressollette E, Ragot S, Bouleti C, Christiaens LP. Optical Coherence Tomography to Better Assess Chronic Total Occlusion Percutaneous Intervention Results: The PERFECTO Study. JACC Adv. 2025 Oct;4(10 Pt 2):102125. doi: 10.1016/j.jacadv.2025.102125. Epub 2025 Sep 9. PMID 40930013